CLINICAL TRIAL: NCT04751162
Title: An Observational Study To Monitor Lung Cancer Patients Activity And Assess Performance Status Through A Wearable Device.
Brief Title: A Study To Monitor Lung Cancer Patients Activity And Assess Performance Status Through A Wearable Device.
Acronym: Lupa-01
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML42283
Record Dates: First submitted 2021-01-12; First posted 2021-02-11 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Phase I: Participants will be asked to wear an actigraphy device (wearable) and to install a mobile application on their smartphones for tracking PA, SQ and symptoms for 3 weeks The ECOG-PS will be assessed by clinician at both, baseline and subsequent visit after the 3 weeks.
  Interventions: Device: Actigraphy device (wearable) and mobile application
- Phase II: Participants will be equipped with both devices (wearable and mobile application) for further monitoring during the following 9 weeks. Study participants will undergo scheduled visits according to local standard practice. The study will progress to Phase II just in case any of the following conditions are met at the end of Phase I:
  * The average time of use of the wearable device is equal or over 96 hours/week/participant, OR
  * The average SUS score is equal or above 68, OR
  * The average adherence to the app is equal or above 80%, measured as the rate of submitted ePROMs through the app.
  Interventions: Device: Actigraphy device (wearable) and mobile application

INTERVENTIONS:
Device: Actigraphy device (wearable) and mobile application — Participants will be asked to wear an actigraphy device (wearable) and to install a mobile application on their smartphones (cf. Broderick et al., 2019) for tracking PA, SQ and symptoms for 3 weeks

SUMMARY:
The current research is a non-interventional (NIS) study seeking to support objective Performance Status (PS) assessments in the particular context of metastatic NSCLC adult patients. To do so, the study comprises two phases. Phase I addresses a feasibility mixed-methods (quantitative-qualitative) approach. It primarily focuses on examining perceived technology usability in a limited sample of participants and feasibility of translating the actigraph data into PS scores (focus expert group). Phase II focuses on to primarily examine associations between technology collected data and ECOG-PS in a larger sample of participants.

ELIGIBILITY:
Inclusion Criteria

Participants must meet the following criteria for study entry:

* 18 or more years of age.
* Able to understand and provide the study informed consent.
* Able to demonstrate basic digital literacy (e.g. knows how to communicate through instant messaging apps or similar).
* ECOG PS of 0, 1 or 2 assessed by physician.
* Life expectancy ≥ 12 weeks
* Histopathologically or cytologically confirmed Non-small cell lung cancer (NSCLC) according to the International Association for the Study of Lung Cancer (IASLC) histopathological classification. Mixed or combined subtypes with component of small cell lung cancer according to the IASLC are not allowed.
* Metastatic NSCLC participants.
* Able to receive 1st line specific antitumor therapy defined by local practice and decision of attended oncologist.

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from study entry:

* Any medical or social condition deemed by the investigator to be likely to interfere with a participant's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
* Participants with advanced LC and a known sensitizing driver mutation: activating EGFR mutation, ALK gene rearrangement, ROS1+ gen rearrangement, BRAF mutation.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures.

Uncontrolled tumor-related pain. Participants requiring pain medication must be on a stable regimen at study entry. Symptomatic lesions amenable to palliative radiotherapy (e.g., bone metastases or metastasis causing nerve impingement) should be treated prior to enrollment. Asymptomatic metastatic lesions whose further growth would likely cause functional deficits or intractable pain (e.g., epidural metastasis that is not presently associated with spinal cord compression) should be considered for locoregional therapy if appropriate prior to enrollment.

* Pregnant or breastfeeding woman.
* Leptomeningeal disease.
* Participants with any of the following central nervous system (CNS) metastases:

  * Symptomatic CNS metastases with need of increasing doses of corticosteroids.
  * Carcinomatous meningitis.
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for ≥ 2 weeks prior to study entry.
* Oncological history:
* Have a previous or concurrent cancer that is distinct in primary (non-pulmonary) site or histology, except carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta and Tis [carcinoma in situ]) or any previous cancer curatively treated with last specific treatment more than 3 years ago without evidence of recurrence.
* Malignancies other than NSCLC within 5 years prior to randomization, with the exception of those with a negligible risk of metastasis or death and treated with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated with curative intent, or ductal carcinoma in situ treated surgically with curative intent).

Severe cardiovascular and pulmonary disease (e.g. myocardial infarction, unstable angina pectoris, coronary angioplasty or stenting, deep vein thrombosis, stroke, pulmonary fibrosis, active uncontrolled bleeding, or a known bleeding diathesis) less than 6 months before inclusion. New York Heart Association Class III or IV congestive heart failure, ventricular arrhythmias, or uncontrolled blood pressure.

* Any psychiatric diagnosis.
* Observed cognitive impairment or disease with cognitive impairment such as Alzheimer's Disease or Parkinson's Disease
* Severe infections within 4 weeks prior to randomization including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Major surgical procedure within 4 weeks prior to randomization or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
* Inability to understand the local language.
* Allergic to dedicated wearable material.
* Currently enrolled in a Clinical Trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First line metastatic NSCLC Patients
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
ECOG-PS assessment of LC participants measured by clinical investigators | From baseline up to 9 months
  ECOG-PS: Eastern Cooperative Oncology Group Performance Status (Oken et al., 1982)
ECOG-PS assessment of LC participants measured by data collected through wearable and a mobile application | From baseline up to 9 months
  ECOG-PS: Eastern Cooperative Oncology Group Performance Status (Oken et al., 1982)
Usability of the mobile application perceived by clinical investigators | From baseline up to 9 months
  System Usability: SUS questionnaire (Brooke, 1986) and usability questionnaire adapted from (Kim et al., 2017). This is a 10-item scale based on a 5-point Likert response measuring strength and agreement of usability. Total scores range from 0 to 100 with score = 68 considered acceptable usability.
Usability of the mobile application perceived by LC participants | From baseline up to 9 months
  System Usability: SUS questionnaire (Brooke, 1986) and usability questionnaire adapted from (Kim et al., 2017). This is a 10-item scale based on a 5-point Likert response measuring strength and agreement of usability. Total scores range from 0 to 100 with score = 68 considered acceptable usability.
Usability of the wearable device perceived by LC participants | From baseline up to 9 months
  System Usability: SUS questionnaire (Brooke, 1986) and usability questionnaire adapted from (Kim et al., 2017). This is a 10-item scale based on a 5-point Likert response measuring strength and agreement of usability. Total scores range from 0 to 100 with score = 68 considered acceptable usability.
Usability of the wearable device perceived by clinical investigators | From baseline up to 9 months
  System Usability: SUS questionnaire (Brooke, 1986) and usability questionnaire adapted from (Kim et al., 2017). This is a 10-item scale based on a 5-point Likert response measuring strength and agreement of usability. Total scores range from 0 to 100 with score = 68 considered acceptable usability.

SECONDARY OUTCOMES:
Sensitivity to changes in ECOG-PS over time measured by clinical investigators | From baseline up to 9 months
  ECOG-PS: Eastern Cooperative Oncology Group Performance Status (Oken et al., 1982)
Sensitivity to changes in ECOG-PS over time measured by wearable and mobile application | From baseline up to 9 months
  ECOG-PS: Eastern Cooperative Oncology Group Performance Status (Oken et al., 1982)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- Spain (10):
  - Fundacion Hospital de Alcorcon, Alcorcón, Madrid
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta; Departamento de Oncologia Medica, Girona
  - Hospital Universitario Clínico San Cecilio; Servicio de oncologia, Granada
  - Hospital 12 de Octubre; Servicio de Digestivo, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Hospital Universitario Virgen del Rocio; Servicio de Oncologia, Seville
  - Hospital Sant Pau i Santa Tecla; Servicio de Oncologia, Tarragona
  - Hospital Universitario la Fe; Servicio de Oncologia, Valencia